CLINICAL TRIAL: NCT05199974
Title: ( Comparison Between ) Conventional and Modified Smead Jones Method for Abdominal Mass Closure in Emergency Midline Laparotomy
Brief Title: Comparison Between Conventional and Modified Smead Jones Method for Mass Closure in Emergency Midline Laparotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Adham Kadry Metawee, resident doctor at general surgery department sohag university hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: soh-med-21-12-08
Record Dates: First submitted 2021-12-13; First posted 2022-01-20 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Midline Laparotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Linea alba was closed with conventional continuous technique . (Active Comparator): Group A: 25 patients included . Linea alba will be closed with conventional continuous technique .
  Interventions: Procedure: Midline abdominal closure
- Group B: Linea alba was closed with Modified Smead Jones technique with Far-near near-far technique. (Active Comparator): Group B:25 patients included. Linea alba will be closed with Modified Smead jones technique with Far-near near-far technique.
  Interventions: Procedure: Midline abdominal closure

INTERVENTIONS:
Procedure: Midline abdominal closure — Abdominal Closure in Emergency Midline Laparotomy

SUMMARY:
The occurrence of sudden disruption of abdominal wall laparotomy wound is a major disaster and a major psychological trauma to the patient . Acute wound dehiscence is defined as postoperative separation of the abdominal musculoaponeurotic layers within 30 days after operation.

Many risk factors were incriminated in causation of burst abdomen including malnutrition, anemia, hypo-proteinemia, pre and post-operative prolonged steroid therapy, peritonitis, malignancy, jaundice, uremia and post-operative abdominal distension or cough.

Wound dehiscence may be related to the technique of closure of abdomen and the sutures used. Numerous studies have been conducted evaluating many closure techniques and suture materials.

There is a number of studies evaluating various closure techniques and suture materials to prevent wound dehiscence following emergency midline laparotomy. In developing countries such as India, most patients operated as an emergency develop wound dehiscence such as they have prolonged intraperitoneal sepsis and malnutrition.

The current opinion for closure of a midline incision is mass closure with non-absorbable or slowly absorbable suture . Tension is distributed evenly along the length of the wound.

The standard technique for abdominal closure is 'mass closure' (closing all layers of the abdominal wall, excluding the skin), usually with nonabsorbable sutures, although 'slow-resorbing' sutures such as polydioxanone (PDS) are also widely used .

In Smead-Jones method of closure tension between two loops is distributed in such a way that the fascial edges are well approximated. Originally described method was interrupted. Continuous method has advantage of being faster and has less risk of wound dehiscence due to dynamic distribution of increased tension in postoperative period due to see-saw effect. We proposed modification of original Smead-Jones technique by doing it in continuous manner to increase the benefits and found this method to be fast, cost-effective, equally effective in controlling wound infection and better than interrupted technique to prevent wound dehiscence.

ELIGIBILITY:
Inclusion Criteria:

* Any patient has risk factor for weak scar who underwent emergency laparotomy through midline incision .

Exclusion Criteria:

* Patients who had previous laparotomy.
* patients who underwent laparotomy through incisions other than midline incisions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Number of burst abdomen post operative | 1 month
  Number of burst abdomen postoperative in emergency midline laparotomy

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sajid MS, Parampalli U, Baig MK, McFall MR. A systematic review on the effectiveness of slowly-absorbable versus non-absorbable sutures for abdominal fascial closure following laparotomy. Int J Surg. 2011;9(8):615-25. doi: 10.1016/j.ijsu.2011.09.006. Epub 2011 Oct 30. PMID 22061310
- [Background] Begum B, Zaman R, Ahmed M, Ali S. Burst abdomen-A preventable morbidity. Mymensingh Med J. 2008 Jan;17(1):63-6. PMID 18285735
- [Background] Rucinski J, Margolis M, Panagopoulos G, Wise L. Closure of the abdominal midline fascia: meta-analysis delineates the optimal technique. Am Surg. 2001 May;67(5):421-6. PMID 11379640